CLINICAL TRIAL: NCT02568644
Title: Double-blind Placebo-controlled Clinical Trial of Ginger (Zingiber Officinale) Addition to Ketoprofen for the Acute Treatment of Migraine Attacks
Brief Title: Ginger Capsules for the Acute Treatment of Migraine Attacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Antonio L Teixeira Jr, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE 21057913.9.0000.5135
Record Dates: First submitted 2015-10-02; First posted 2015-10-06 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Migraine
Keywords: Migraine; Ginger; Acute treatment
MeSH Terms: conditions — Migraine Disorders | interventions — Phytotherapy; Cellulose; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extract of ginger (Experimental): People (both genders) who went to the emergency room of the Hospital Vera Cruz (Belo Horizonte, MG, BR) with a migraine attack received two capsules of ginger extract (containing 5% of gingerols) and intravenous ketoprofen (100mg).
  Interventions: Dietary Supplement: Extract of ginger; Drug: Intravenous ketoprofen
- Cellulose (Placebo Comparator): People (both genders) who went to the emergency room of the Hospital Vera Cruz (Belo Horizonte, MG, BR) with a migraine attack received two placebo capsules (cellulose) and intravenous ketoprofen (100mg).
  Interventions: Other: Cellulose; Drug: Intravenous ketoprofen

INTERVENTIONS:
Dietary Supplement: Extract of ginger — People (both genders) who went to the emergency room of the Hospital Vera Cruz (Belo Horizonte, MG, BR) with a migraine attack received two capsules of ginger extract (containing 5% of gingerols).
  Other Names: Phytotherapy
  Arms: Extract of ginger
Other: Cellulose — People (both genders) who went to the emergency room of the Hospital Vera Cruz (Belo Horizonte, MG, BR) with a migraine attack received two placebo capsules (cellulose).
  Other Names: Placebo
  Arms: Cellulose
Drug: Intravenous ketoprofen — People (both genders) who went to the emergency room of the Hospital Vera Cruz (Belo Horizonte, MG, BR) with a migraine attack received intravenous ketoprofen (100mg).
  Other Names: Nonsteroidal anti-inflammatory drug

SUMMARY:
The main objective of the study was to evaluate ginger efficacy as an adjuvant to ketoprofen for the treatment of headache and other symptoms related with migraine attacks.

DETAILED DESCRIPTION:
Patients with the diagnosis of migraine according to the International Headache Society (IHS) criteria were enrolled in the study during a migraine attack. Patients received two 200 mg capsules of dry ginger extract (5% active ingredient) or two capsules of placebo (cellulose) in addition to an intravenous dose of ketoprofen (100 milligrams - mg) to treat the migraine attack.

ELIGIBILITY:
* Inclusion Criteria:

  * Migraine diagnosis for at least one year;
  * Migraine attack with moderate or severe pain intensity;
  * One to six migraine attacks per month.
* Exclusion Criteria:

  * Patients with headaches not characterized as migraine;
  * Pregnant or lactating women;
  * Fertile and sexually active women who do not use contraception;
  * Abuse of painkillers, alcohol or drugs;
  * People with hypersensitivity to ginger;
  * People with other neurological diseases;
  * People in use of anticoagulant drugs;
  * People who have started the disease after 50 years old.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adaliene VM Ferreira, PhD, Study Director — Federal University of Minas Gerais; Laís B Martins, Ma, Study Chair — Federal University of Minas Gerais; Antônio L Teixeira, PhD, Principal Investigator — Federal University of Minas Gerais

REFERENCES:
- [Derived] Martins LB, Rodrigues AMDS, Rodrigues DF, Dos Santos LC, Teixeira AL, Ferreira AVM. Double-blind placebo-controlled randomized clinical trial of ginger ( Zingiber officinale Rosc.) addition in migraine acute treatment. Cephalalgia. 2019 Jan;39(1):68-76. doi: 10.1177/0333102418776016. Epub 2018 May 16. PMID 29768938

RESULTS

PARTICIPANT FLOW:
Groups:
- Extract of Ginger: 30 people (both genders) who went to the emergency room of the Hospital Vera Cruz (Belo Horizonte, MG, BR) with a migraine attack received two capsules of ginger extract (containing 5% of gingerois) and intravenous ketoprofen (100mg).
  Extract of ginger: 30 people (both genders) who went to the emergency room of the Hospital Vera Cruz (Belo Horizonte, MG, BR) with a migraine attack received two capsules of ginger extract (containing 5% of gingerois).
  Intravenous ketoprofen: 30 people (both genders) who went to the emergency room of the Hospital Vera Cruz (Belo Horizonte, MG, BR) with a migraine attack received intravenous ketoprofen (100mg).
- Cellulose: 30 people (both genders) who went to the emergency room of the Hospital Vera Cruz (Belo Horizonte, MG, BR) with a migraine attack received two placebo capsules (cellulose) and intravenous ketoprofen (100mg).
  Cellulose: 30 people (both genders) who went to the emergency room of the Hospital Vera Cruz (Belo Horizonte, MG, BR) with a migraine attack received two placebo capsules (cellulose).
  Intravenous ketoprofen: 30 people (both genders) who went to the emergency room of the Hospital Vera Cruz (Belo Horizonte, MG, BR) with a migraine attack received intravenous ketoprofen (100mg).
Period: Overall Study
Arm/Group | Extract of Ginger | Cellulose
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extract of Ginger | Cellulose | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (8.8) | 34.3 (9.1) | 33.5 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Marital Status [Count of Participants; unit: Participants] — Marital status was classified:
  Married [n (%)] Single [n (%)] Widowed/Divorced [n (%)]
  Participants
    Single | 17 | 15 | 32
    Widowed/Divorced | 1 | 2 | 3
    Married | 12 | 13 | 25
Occupation [Count of Participants; unit: Participants] — Work [n (%)] Do not work [n (%)]
  Participants
    Work | 30 | 25 | 55
    Do not work | 0 | 5 | 5
Migraine Diagnosis [Count of Participants; unit: Participants] — M. with aura [n (%)] M. without aura [n (%)]
  Participants
    Migraine with aura | 15 | 12 | 27
    Migraine without aura | 15 | 18 | 33
Length of disease [Mean (Standard Deviation); unit: years] | 11.0 (10.7) | 10.0 (9.6) | 10.5 (10.1)
Age of onset the disease [Mean (Standard Deviation); unit: years] | 21.0 (9.8) | 23.1 (9.4) | 22.7 (9.6)
Number of migraine attacks/month [Mean (Standard Deviation); unit: migraine attacks/month] | 2.2 (1.3) | 2.7 (1.2) | 2.4 (1.2)
Migraine Disability Test (MIDAS) [Mean (Standard Deviation); unit: units on a scale] — Migraine Disability Test (MIDAS)
  The MIDAS is a questionnaire designed to quantify headache-related disability over a 3 month period.
  Total Score is obtained with the sum of days lost in social, domestic and work activities
  The total score corresponding to four categories:
  0 to 5 = Grade I - Llittle or no disability 6 to 10 = Grade II - Mild disability 11 to 20 = Grade III - Moderate disability 21 or + = Grade IV - Severe disability
  units on a scale | 17.4 (14.2) | 14.2 (8.3) | 15.8 (11.2)
Headache Impact Test, version 6 (HIT-6) [Mean (Standard Deviation); unit: units on a scale] — Headache Impact Test, version 6 (HIT-6)
  HIT-6 measures the disability caused by headaches in the previous month. This questionnaire consists of six questions whose answer alternatives are given in frequency. The result is the sum of the points for each answer.
  The four headache impact severity categories are little or no impact (49 or less), some impact (50-55), substantial impact (56-59), and severe impact (60-78).
  units on a scale | 64.6 (5.5) | 66.9 (4.2) | 65.7 (4.8)
BDI [Mean (Standard Deviation); unit: units on a scale] — Beck Depression Inventory
  The BDI measures the severity of depressive episodes. It is a self-report questionnaire with 21 groups of statements that express levels of severity of depressive symptoms ranging from 0 to 3 points.
  The standard cut-off scores are as follows:
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-+: indicates severe depression.
  units on a scale | 11.2 (6.8) | 13.9 (9.3) | 12.5 (8.0)
Pain intensity (Four-point Scale) [Mean (Standard Deviation); unit: units on a scale] — The 4-point verbal scale consists of pain classification in scores between zero and three that correspond to: 0 - Absence of pain, 1 - Mild Pain, 2 - Moderate Pain and 3 - Severe pain
  units on a scale | 2.46 (0.09) | 2.56 (0.09) | 2.51 (0.09)
Pain intensity (Faces Pain Scale) [Mean (Standard Deviation); unit: units on a scale] | 2.90 (0.17) | 2.96 (0.17) | 2.93 (0.17)
Pain intensity (Visual Numeric Scale) [Mean (Standard Deviation); unit: units on a scale] — The numerical visual scale has a score ranging from zero to 10 and is associated with the description of pain intensity and functional capacity, where zero corresponds to absence of pain and ten to maximum, disabling pain.
  units on a scale | 7.03 (0.26) | 7.63 (0.25) | 7.33 (0.25)

OUTCOME MEASURES:

1. Primary Outcome: Change in Headache Severity.
Description: The severity of headache was assessed with four-point scale. Scale ranges: 0 - Absence of pain, 1 - Mild Pain, 2 - Moderate Pain and 3 - Severe pain Higher scores mean a worse outcome
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extract of Ginger | Cellulose
Number analyzed (Participants) | 30 | 30
units on a scale | 0.81 (0.04) | 0.97 (0.07)

2. Primary Outcome: Change in Headache Severity.
Description: The severity of headache was assessed with visual numeric scale. Scale ranges: from zero (absence of pain) to 10 (maximum intensity of pain). Higher scores mean a worse outcome.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extract of Ginger | Cellulose
Number analyzed (Participants) | 30 | 30
units on a scale | 1.03 (0.29) | 2.30 (0.46)

3. Primary Outcome: Change in Headache Severity.
Description: The severity of headache was assessed with faces pain scale. It is a self-reported pain scale consisting of face drawings which have a score ranging from zero (absence of pain) to five (maximal intensity of pain).
  Higher scores mean a worse outcome.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extract of Ginger | Cellulose
Number analyzed (Participants) | 30 | 30
units on a scale | 0.43 (0.13) | 0.90 (0.18)

4. Secondary Outcome: Change in Serum Levels of Biomarkers.
Description: Evaluated biomarkers: neurotrophic factors and inflammatory mediators.
Time Frame: 2 hours
Population: Brain derived neurotrophic factor - BDNF (pg/mL)
Measure: Median (95% Confidence Interval); unit: BDNF (pg/mL)
Groups:
- Extract of Ginger: People (both genders) who went to the emergency room of the Hospital Vera Cruz (Belo Horizonte, MG, BR) with a migraine attack received two capsules of ginger extract (containing 5% of gingerois) and intravenous ketoprofen (100mg).
  Extract of ginger: People (both genders) who went to the emergency room of the Hospital Vera Cruz (Belo Horizonte, MG, BR) with a migraine attack received two capsules of ginger extract (containing 5% of gingerois).
  Intravenous ketoprofen: People (both genders) who went to the emergency room of the Hospital Vera Cruz (Belo Horizonte, MG, BR) with a migraine attack received intravenous ketoprofen (100mg).
Arm/Group | Extract of Ginger | Cellulose
Number analyzed (Participants) | 30 | 30
BDNF (pg/mL) | 6077 [5694 to 6944] | 6503 [5929 to 7244]

ADVERSE EVENTS:
Arm/Group | Extract of Ginger | Cellulose
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 3/30 | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Extract of Ginger (N=30) | Cellulose (N=30)
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Dizziness (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes